CLINICAL TRIAL: NCT00690690
Title: No Excuses/Sin Buscar Excusas Intervention to Reduce Latino Men's HIV Risks
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: Education Development Center, Inc. (Industry); Callen-Lorde Community Health Center (Other); Hispanic AIDS Forum, Inc. (Industry)
Responsible Party: Education Development Center, Inc., Lydia O'Donnell
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CDC-NCHHSTP-5142
Record Dates: First submitted 2008-06-03; First posted 2008-06-05 (Estimated); Last update posted 2010-03-09 (Estimated); Status verified 2010-03

CONDITIONS: HIV Infections
Keywords: HIV Seronegativity; HIV risk behavior; Unprotected sex; men who have sex with men; gay; Latino; unsafe sex; high risk sex
MeSH Terms: conditions — HIV Infections; Unsafe Sex; Homosexuality | interventions — Videotape Recording

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- video (Experimental)
  Interventions: Behavioral: Video (group-delivered video-based intervention)
- HCT (Active Comparator): Offer of HIV counseling and testing
  Interventions: Behavioral: HCT

INTERVENTIONS:
Behavioral: Video (group-delivered video-based intervention) — group-delivered video-based intervention
  Arms: video
Behavioral: HCT — Offer of HIV counseling and testing
  Arms: HCT

SUMMARY:
The overall goal of this study is to develop and evaluate a brief, video-based, group-level intervention designed to reduce sexual risk taking among culturally diverse English- and Spanish-speaking Latino men who have sex with men (MSM).

ELIGIBILITY:
Inclusion Criteria:

* Be between the ages of 18 - 49
* Self-identify as Latino or Hispanic
* Speak English and/or Spanish
* Reside in NYC and not plan to move in the next 3 months
* Have had 2 or more sex partners in the last 3 months
* Have had at least 1 male sex partner in the last 3 months
* Have engaged in unprotected anal intercourse with at least one male partner in the last 3 months
* Be HIV negative or not know their status

Exclusion Criteria:

* Participated in a program (research or non-research) during the past 6 months where they have received HIV prevention education (e.g. an in-person or online group session, workshop, support group).
* Report being HIV-positive

Ages: 18 Years to 49 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 370 (Actual)
Dates: Start 2008-06; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Sexual risk behavior | past 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Lydia O'Donnell, PhD, Principal Investigator — Education Development Center, Inc.
Locations (1):
- Education Development Center, Inc., New York, New York, United States